CLINICAL TRIAL: NCT01461382
Title: Workplace Intervention: Activity Monitoring as a Tool for Corporate Wellness and Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James Levine, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 07-003809
Record Dates: First submitted 2011-10-24; First posted 2011-10-28 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I (Experimental): Entered Study May 2008.
  Interventions: Other: Treadmill Desks
- Phase II (Experimental): Phase II entered 6 months after Phase I. Phase II was a no intervention control for 6 months, then followed an identical intervention protocol to Phase I.
  Interventions: Other: Treadmill Desks

INTERVENTIONS:
Other: Treadmill Desks — Treadmill Desk were installed in subjects personal workspace.
  Arms: Phase I
Other: Treadmill Desks — Treadmill desks were installed in subjects personal workspace six months after phase I started.
  Arms: Phase II

SUMMARY:
Is a one-year intervention with Treadmill Desks associated with increased employee daily physical activity and decreased sedentariness.

36 employees with sedentary jobs (87 + 27 kg, BMI 29 + 7 kg/m2) used a Treadmill Desk for one year. Daily Physical Activity, work performance, body composition, and blood variables were measured at Baseline and 6 and 12 months after the Treadmill Desk intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited regardless of race/ethnicity.

Exclusion Criteria:

* Definite termination criteria.

  * Request by subject to leave study.
  * Evidence of deliberate non-compliance (e.g.; placing activity instruments on another individual, deliberate destruction of instruments).
  * Pregnancy.
  * Alcohol abuse; elicit drug abuse.
  * Development of chronic condition that is likely to impact on metabolic variables or requiring medications likely to impact on metabolic variables or likely to result in subject being unable to participate (e.g., Grave's disease, hypothyroidism, rheumatoid arthritis requiring steroids or limiting mobility, congestive cardiac failure, neurological disorder such as multiple sclerosis or stroke).
  * Development of acute condition that is likely to impact on metabolic variables or requiring medications likely to impact on metabolic variables or likely to result in subject being unable to participate (e.g., motor vehicle accident with multiple fractures, myocardial infarction, major depression).

Potential termination criteria.

Development of acute or chronic condition that may impact on metabolic variables or requiring medications likely to impact on metabolic variables or likely to result in subject being unable to participate. Subjects will be reviewed on a subject-by-subject basis and will be reported to the Safety-Monitoring Panel. Specific action plans are pre-assigned for:

* Diabetes (two fasting plasma glucose values >126 mg/dl). Here, glycosylated hemoglobin will be measured three monthly (by the study) and subjects referred to their local physician for preventative screening. Subjects will be excluded from further study with any glycosylated hemoglobin value of >8% or symptomatic hyperglycemia.
* Depression or low mood. Here, all patients will be asked to be evaluated by their primary care physician and if appropriate referred to a psychiatrist. The opinion of the psychiatrist will be used to determine continuance or termination in the protocol.

This does not represent a comprehensive listing of criteria or causes. All subjects who withdraw or whom are withdrawn from the study or whom are considering/being considered for withdrawal will be referred to the Safety-Monitoring Panel. These subjects' data will be scrutinized (whether terminated or not) separately to assess for association of intervention with a specific adverse outcome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Daily Physical Activity | 1 year
  Measured for all waking hours using tri-axial accelerometry.

SECONDARY OUTCOMES:
Body Weight | baseline, 6 months, 12 months
Body Composition | baseline, 6 months, 12 months
Venous blood | baseline, 6 months, 12 months
Work performance | baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James A Levine, MD PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States